CLINICAL TRIAL: NCT00195754
Title: The Safety of Divalproex Sodium Extended Release Tablets in Migraine Prophylaxis: An Open-Label Extension Study in Adolescents
Brief Title: A Phase III Open-Label, Multi-Center, Long-Term Extension Study of Depakote ER in Subjects Who Either Completed or Prematurely Discontinued Due to Ineffectiveness From Study M02-488.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-554
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Migraines
Keywords: Migraines; Depakote ER; divalproex sodium
MeSH Terms: conditions — Migraine Disorders | interventions — Valproic Acid

INTERVENTIONS:
Drug: divalproex sodium

SUMMARY:
The purpose of this study is to determine if long-term treatment, up to 1 year, with Depakote ER is safe in the reduction of occurrence of migraine headaches in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subject and subject's legal representative have voluntarily signed and dated an IRB-approved informed assent form and an IRB-approved informed consent form, respectively, before any study-specific procedures or tests are performed;
* The subject was randomized into Study M02-488 and either completed the study or prematurely discontinued due to ineffectiveness; and
* The subject is male or non-pregnant, non-lactating female

Exclusion Criteria

* Female, of childbearing potential, and not using an effective method of birth control (e.g., total sexual abstinence or contraceptives).
* Experienced a serious adverse event in Study M02-488 which the investigator considered "possibly" or "probably related" to study drug; or
* In the investigator's opinion, long-term treatment with Depakote ER for migraine prophylaxis is contraindicated.
* For any reason, subject is considered by the investigator to be an unsuitable candidate to receive divalproex sodium or to participate in this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2004-07

PRIMARY OUTCOMES:
Safety outcome measure | 12 months

SECONDARY OUTCOMES:
Migraine headache rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 800-633-9110, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States